CLINICAL TRIAL: NCT07274280
Title: Comparative Evaluation of Ambu AuraGain, LarySeal Pro LMA and I-gel in Pediatric Airway Management for Day-Case Surgery Under Controlled Ventilation: A Randomized Comparative Trial
Brief Title: Comparative Evaluation of Ambu AuraGain, LarySeal Pro and I-gel in Pediatric Airway Management for Day-Case Surgery Under Controlled Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Emad Mohamed Ahmed Abdelhafez, Lecturer of Anesthesia, Surgical Intensive Care and Pain Management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: N-288-2025
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Airway Control

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: Ambu AuraGain LMA (Active Comparator): supraglottic Airway device used for airway control
  Interventions: Device: supraglottic airway device
- Group II: LarySeal Pro LMA (Active Comparator): supraglottic airway device used for airway control
  Interventions: Device: supraglottic airway device
- Group III: I-gel (Active Comparator): supraglottic airway device used for airway control
  Interventions: Device: supraglottic airway device

INTERVENTIONS:
Device: supraglottic airway device — use of supraglottic airway device as an airway control device for pediatric patients during day case surgery under controlled ventilation

SUMMARY:
This study aims to compare the Ambu AuraGain, LarySeal Pro LMA, and i-gel regarding their insertion characteristics, ventilation efficacy, risk of gastric insufflation, fiberoptic view quality, intraoperative and postoperative airway-related complications, and hemodynamic stability.165 consecutive pediatric patients aged 2-9 years, weighing 10-30 kg, American Society of Anesthesiologists (ASA) physical status I or II, and scheduled for elective day-case surgery suitable for supraglottic airway device (SGAD) use.Patients will be randomly assigned (n= 55 per group) using a computer-generated random number sequence (www.random.org) to one of three groups:

* Group I: Ambu® AuraGain TM (Ambu Ltd Xiang Yu Xiamen, Fujian, China)
* Group II: LarySeal Pro® LMA (Flexicare Medical Limited, Cynon Valley Business Park, Mountain Ash, UK).Patients will receive oral midazolam before anesthesia, followed by standard monitoring, induction with sevoflurane, fentanyl, and atracurium, and insertion of an appropriately sized SGAD by experienced anesthesiologists. Ventilation quality, oropharyngeal leak pressure (OLP), peak airway pressure (Ppeak), fiberoptic glottic view, and gastric insufflation by ultrasound will be assessed. Anesthesia will be maintained with controlled ventilation and cuff pressure adjusted to 60 cmH₂O. At the end, neuromuscular blockade will be reversed, devices removed upon awakening, and patients observed for complications such as laryngospasm, Outcome parameter (s):
* Oropharyngeal Leak Pressure (OLP).
* Demographic and Clinical Data.
* Hemodynamics.
* Insertion Data.
* Peak Airway Pressure (Ppeak).
* Fiberoptic Glottic View Assessment.
* Ultrasound Assessment of Gastric Insufflation.
* Perioperative Complications.bronchospasm, or sore throat.
* Group III: I-gelTM (Intersurgical Ltd, Berkshire, RG41 2RZ, UK).

ELIGIBILITY:
Inclusion Criteria:

* • Age 2-9 years.

  * Weight 10-30 kg.
  * ASA Physical Status I or II.
  * Elective day-case surgery requiring general anesthesia with controlled ventilation using an SGAD.
  * Written informed consent from parent(s) or legal guardian(s).

Exclusion Criteria:

* • ASA Physical Status III or IV.

  * Known or predicted difficult airway.
  * History of significant respiratory disease (e.g., asthma requiring frequent medication, active upper respiratory tract infection, reactive airway disease within the past month).
  * History of significant gastroesophageal reflux, hiatal hernia, BMI ≥ 35, or other conditions predisposing to increased aspiration risk.
  * Neuromuscular disorders affecting airway patency or respiratory function.
  * Known allergy or contraindication to study devices or anesthetic medications.
  * Participation in other clinical trials that could influence study outcomes.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal Leak Pressure (OLP) | from enrollment to the end of the study at 6 months

SECONDARY OUTCOMES:
Peak Airway Pressure (P peak) | From enrollement to the end of the study at 6 months
Fiberoptic glottic airway view | From enrollment to the end of the study at 6 months
Ultrasound Assessment of Gastric Insufflation | From enrollement to the end of the study at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- KasrAlainy Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Demographic and clinical data Insertion data of the SGAD (time, successfulness) OLP Ppeak Hemodynamic data Fiberoptic glottic view data Ultrasound assessment of gastric insufflation data Perioperative complication data
Supporting Information: Study Protocol, SAP
Time Frame: January 2025 - january 2026

REFERENCES:
- See also: educational and academic web page — http://www.cu.edu.eg